CLINICAL TRIAL: NCT06275373
Title: The Effect of Teprotumumab on Thyroid Eye Disease and Thyroid Dysfunction
Acronym: Teprotumumab
Status: Recruiting | Type: Observational
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thanh Hoang, Endocrinologist, Walter Reed National Military Medical Center
Other Study IDs: 20-10974
Record Dates: First submitted 2024-01-22; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Thyroid Eye Disease; Graves Ophthalmopathy; Graves Disease
Keywords: Thyroid eye disease; Graves ophthalmopathy; Graves disease
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease | interventions — teprotumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Teprotumumab Injection [Tepezza] — IGF1 monoclonal antibody
  Other Names: Tepezza TM

SUMMARY:
This protocol studies the clinical outcome of patients with active thyroid disease with visually significant signs and symptoms of proptosis, pain, diplopiam lid/orbital edema, or lid/orbital erythema recommended for treatment with teprotumumab infusion (Tepezza®). Patients recommended for treatment will be evaluated by an oculoplastic surgeon (Dr. Eva Chou) and endocrinologist (Dr. Thanh Hoang).

DETAILED DESCRIPTION:
Thyroid eye disease (TED), also known as Graves' orbitopathy or thyroid-associated ophthalmopathy is a rare debilitating autoimmune condition in which immune cells attack the eye muscles and connective tissues within the eye socket, leading to proptosis, pain, diplopia, periorbital and orbital erythema and edema, exposure keratopathy and lagophthalmos, decreased vision, and compressive optic neuropathy. It has an incidence of 1.9 cases per 10,000 population per year. Approximately 25% of patients with autoimmune thyroid disease develop TED within 18 months of diagnosis. Severe optic neuropathy will affect 10% of patients with TED, leading to irreversible vision loss.

The natural history of TED involves an initial active phase, during which the autoimmune process causes the above mentioned morbidity, followed by a quiescent phase. The active period usually lasts 2-3 years and requires monitoring until the disease is quiescent. Until now, treatment during the active period focuses on preserving sight and providing treatment for double vision. Emergent orbital decompression or radiation treatment is reserved for compressive optic neuropathy. Alternative therapies, such as glucocorticoids, have little effect on proptosis and can have dose-limiting side effects. When the active phase "burns" out, the treatment for thyroid eye disease involves rehabilitative surgeries for orbital decompression, followed by strabismus surgery, followed by eyelid recession surgery; altogether, this may involve multiple surgeries which don't reverse the damage of the ocular and orbital tissues.

Tepezza®, or teprotumumab, is a fully human monoclonal insulin-like growth factor-1 receptor (IGF-1R) inhibitor antibody which blocks the inflammatory/autoimmune pathophysiology that underlies thyroid eye disease. It is the first FDA-approved medication for the treatment of adults with thyroid eye disease, reversing inflammatory changes of proptosis and diplopia. In clinical trials, 83% of patients receiving teprotumumab demonstrated a greater than 2 mm reduction in proptosis compared to 10% of participants who received placebo (between-group difference, 73% points; 95% CI = 59-88; P<0.001). Teprotumumab had a quick improvement on each outcome, which was evident at the first postbaseline evaluation at week 6, and the results improved during the 24-week treatment period. This therapy could potentially replace surgery for many patients, including those with more advanced disease.

The investigators propose a retrospective observational chart review of a cohort of adults with active TED without compressive optic neuropathy necessitating urgent orbital decompression or radiation who are undergoing treatment with Tepezza®. Inclusion criteria are patients with a clinical diagnosis of autoimmune thyroid disease and moderate-severe TED with clinical activity including symptoms of proptosis, diplopia, orbital pain, lid/orbital edema, or lid/orbital erythema, and with circulating thyroid stimulating or anti-thyroid auto-antibodies present within the last 18 months from the initiation of treatment. Exclusion criteria include patients with a history of compressive optic neuropathy necessitating urgent orbital decompression or external beam radiation, patients with a history of uncontrolled diabetes, uncontrolled inflammatory bowel disease, patients under 18 years old, and patients who are pregnant or trying to become pregnant.

The primary outcome is CAS score improvement and TSI level.

HLA has been associated with Graves disease and TED in different populations. In White patients, C*07:01, DQA1*05:01, DRB1*03, and DQB1*02:01 are associated with GD risk while DRB1*07:01 and DQA1*02:01 may be protective. However, in Asian patients, GD was noted to be mostly associated with B*46:01, *05:01, DRB1*08:02/03, DRB1*16:02, DRB1*14:03, DRB1*04:05, DQB*05:02 and DQB1*03:03, while DRB1*07:01 DRB1*01:01, DRB1*13:02, and DRB1*12:02 are potentially protective. Likewise, HLA-B*38:02, DRB1*16:02, DQA1*01:02, and DQB1*05:02 have been linked to increased TED risk in Asian patients while HLA-B*54:01 may be protective for TED in White patients.

In this study, the investigators analyze the HLA subtypes and correlate these with responders and non-responders to teprotumumab therapy.

ELIGIBILITY:
Inclusion Criteria:

* only DOD beneficiaries
* adult patients 18 years of age or older
* adult patients with proptosis, ocular/orbital pain, diplopia, lid/orbital edema, or lid/orbital erythema associated with autoimmune thyroid disease

Exclusion Criteria:

* Patients with evidence of compressive optic neuropathy necessitating urgent orbital decompression or external beam radiation
* patients with a history of uncontrolled diabetes mellitus
* patients with a history/diagnosis of uncontrolled inflammatory bowel disease
* patients under age 18 years
* patients who are pregnant or trying to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study participants were 18-80 years old at the time of treatment with teprotumumab, diagnosed with autoimmune thyroid disease (positive stimulating thyroid receptor antibodies or elevated TSI), presenting with active eye disease (associated with at least one of the following: lid retraction of ≥2 mm, moderate or severe soft-tissue involvement, proptosis of ≥3 mm above the normal values for race and sex, and periodic or constant diplopia), and treated with at least one dose of teprotumumab.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2026-05-12 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Ophthalmological Clinical Activity Score (CAS) scoring | 6-12 months post treatment
  CAS scoring (1 to 10)
Thyroid stimulating immunoglobulin | 6-12 months post treatment
  TSI (IU/L)

SECONDARY OUTCOMES:
HLA subtypes | 6-12 months
  HLA subtypes

CONTACTS AND LOCATIONS:
Overall Officials: Thanh D Hoang, DO, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No